CLINICAL TRIAL: NCT00908128
Title: A Single-Dose, Replicate, Comparative Bioavailability Study of Two Formulations of Mycophenolate Mofetil 500 mg Tablets Under Fed Conditions
Brief Title: Mycophenolate Mofetil Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2006-1264
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolate Mofetil (test) First (Experimental): Mycophenolate Mofetil Tablets, 500 mg dosed in first period followed by CellCept® Tablets, 500 mg dosed in second period; sequence repeated in third and fourth periods.
  Interventions: Drug: Mycophenolate Mofetil
- CellCept® (reference) First (Active Comparator): CellCept® Tablets, 500 mg dosed in first period followed by Mycophenolate Mofetil Tablets, 500 mg dosed in second period; sequence repeated in third and fourth periods.
  Interventions: Drug: CellCept®

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil 500 mg Tablet
  Arms: Mycophenolate Mofetil (test) First
Drug: CellCept® — CellCept® Tablets, 500 mg
  Arms: CellCept® (reference) First

SUMMARY:
The objective of this study was to evaluate the comparative bioavailability between Mycophenolate Mofetil 500 mg Tablets (test) and CellCept® 500 mg Tablets (reference), after a single-dose in healthy subjects under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male subjects, 18 years of age or older.
* Healthy, non-smoking post-menopausal or surgically sterile females 18 years of age or older.
* BMI ≥ 19 and ≤ 30.
* Negative for:

  1. HIV.
  2. Hepatitis B surface antigen and Hepatitis C antibody.
  3. Using drugs of abuse test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and methadone).
  4. Urine cotinine test
  5. Serum HCG consistent with pregnancy (females only)
* No significant diseases or clinically significant findings in a physical examination.
* No clinically significant abnormal laboratory values.
* No clinically significant findings in vital signs measurements and a 12-lead electrocardiogram (ECG).
* Be informed of the nature of the study and given written consent prior to receiving any study procedure.
* Females who participate in this study must be unable to have children:

  1. post-menopausal for at least 1 year - no menstrual cycle for 12 months and LH and FSH levels judged by a physician to be consistent with post-menopausal status.

     OR
  2. Proof of surgical sterility.
* Females who participate in this study are not pregnant and/or non-lactating.

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition.
* Known or suspected carcinoma.
* Known or suspected increased susceptibility to infection.
* Known history or presence of active tuberculosis (TB).
* Results of a previous TB skin test greater than 5 mm in diameter.
* Lived in or traveled, during the last 8 weeks, to a country defined by the Public Health Agency of Canada as having WHO estimated sputum smear positive pulmonary TB rate of 15 per 100,000 or higher.
* Known history or presence of:

  1. Hypersensitivity or idiosyncratic reaction to mycophenolate mofetil and/or any other drug substances with similar activity.
  2. Alcoholism within the last 12 months.
  3. Drug dependence and/or substance abuse.
  4. Use of tobacco or nicotine-containing products within the last 6 months.
* On a special diet within 4 weeks prior to drug administration (e.g. liquid, protein, raw food diet).
* Participated in another clinical trial or received and investigational product within 30 days prior to drug administration.
* Donated up to 250 mL of blood within the previous 30 days OR Donated from 251 to 499 mL of blood in the previous 45 days OR Donated more than 499 mL of blood in the previous 56 days (based on the Canadian Blood Services guideline for blood donation.
* Females taking oral or transdermal hormonal contraceptives within 14 days preceding period 1 dosing.
* Females having taken implanted or injected hormonal contraceptives within 6 months prior to period 1 dosing.
* Requirement of any non-topical medication (prescription and/or over-the-counter) on a routine basis.
* Difficulty fasting or consuming the standard meals.
* Do not tolerate venipuncture.
* Unable to read or sign the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, MD, PhD., FRCP(C), Principal Investigator — Pharma Medica Research, Inc.
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Period 4
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First
Started | 20 | 19 (One subject withdrew prior to Period 4 dosing due to adverse events)
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil (Test) First | CellCept® (Reference) First | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 18 | 19 | 37
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 9 | 14 | 23
  Black | 4 | 4 | 8
  Asian | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Mycophenolate Mofetil: Mycophenolate Mofetil Tablets, 500 mg dosed in any period.
- CellCept®: CellCept® Tablets, 500 mg dosed in any period.
Arm/Group | Mycophenolate Mofetil | CellCept®
Number analyzed (Participants) | 39 | 39
µg/mL | 7.4578 (3.4339) | 8.2195 (3.9390)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs CellCept®; Test type: Non-Inferiority or Equivalence — Analyses of Variance (PROC MIXED) was performed on lon-transformed AUCt, AUCinf and Cmax parameters; Geometric Test/Ref Ratio x 100 = 90.96, 90% CI [82.40 to 100.41] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | Mycophenolate Mofetil | CellCept®
Number analyzed (Participants) | 39 | 39
µg*hr/mL | 24.5141 (7.3941) | 24.9890 (7.1389)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs CellCept®; Test type: Non-Inferiority or Equivalence — Analyses of Variance (PROC MIXED) was performed on log-transformed AUCt, AUCinf and Cmax parameters; Geometric Test/Ref Ratio x 100 = 99.16, 90% CI [96.24 to 102.16] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of the Last Non-zero Concentration
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | Mycophenolate Mofetil | CellCept®
Number analyzed (Participants) | 39 | 39
µg*hr/mL | 23.3091 (6.9780) | 23.5366 (6.8250)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs CellCept®; Test type: Non-Inferiority or Equivalence — Analyses of Variance (PROC MIXED) was performed on the log-transformed AUCt, AUCinf and Cmax parameters; Geometric Test/Ref Ratio x 100 = 98.78, 90% CI [95.76 to 101.89] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.